CLINICAL TRIAL: NCT02020252
Title: A Pilot Investigation to Examine the Effect of a Multi-Media, Computer Based Tool (Talking Touchscreen) on Enrollment in Adult Oncology-Specific Clinical Trials at an Academic Medical Center
Brief Title: Effect of Multi-Media Tool on Enrollment in Oncology Clinical Trials
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Northwestern University (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB13-1233
Record Dates: First submitted 2013-12-09; First posted 2013-12-24 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer; Gastric Cancer; Pancreatic Cancer
Keywords: clinical trials enrollment; communication; low health literacy; health disparities
MeSH Terms: conditions — Lung Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Touchscreen Participants: New lung, gastric and pancreatic cancer patients presenting to the University of Chicago outpatient oncology clinics, a large research institution located on Chicago's Southside, were identified for study accrual, using the electronic scheduling system.
  Interventions: Behavioral: Testing an interactive technology in a diverse health literary population

INTERVENTIONS:
Behavioral: Testing an interactive technology in a diverse health literary population — Enrollment in therapeutic cancer trials remains low, and is especially challenging for patients with low health literacy. We tested an interactive technology designed for patients with diverse health literacy skills aimed at improving patient receptiveness, willingness, knowledge, self-efficacy and positive attitudes regarding clinical trials.

SUMMARY:
The purpose of this research study is to test a touchscreen computer program, which allows patients to see information on a computer screen regarding cancer care, and specifically clinical trials. The purpose of this research is to help the investigators learn more about how to use technology in the medical setting to improve health outcomes.

DETAILED DESCRIPTION:
Enrollment in therapeutic cancer trials remains low, and is especially challenging for patients with low health literacy. The purpose of this project is to pilot a multi-media technology intervention designed for patients with diverse health literacy skills with the aim of improving patient receptiveness, willingness, knowledge, self-efficacy, and positive attitudes regarding clinical trials. The intervention is comprised of multi-media touchscreen computer program components for clinical trial education and assessment of patient-reported outcomes. Patients presenting for their first oncology appointment were eligible. Patients viewed an interactive teaching video concerning clinical trials that was adapted from the National Institutes of Health. Validated surveys assessing receptiveness, willingness, knowledge, self-efficacy, and positive attitudes regarding clinical trials were administered before and after the test.

ELIGIBILITY:
Inclusion Criteria:

* Adult, English-speaking women and men
* Newly diagnosed with lung, gastric or pancreatic cancer
* Coming to the University of Chicago outpatient oncology clinics for their first oncology visit

There are no Exclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the University of Chicago Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blase Polite, MD, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Polite BN, Cipriano-Steffens TM, Liao C, Miller EL, Arndt NL, Hahn EA. Investigation of a multimedia, computer-based approach to improve knowledge, attitudes, self-efficacy, and receptivity to cancer clinical trials among newly diagnosed patients with diverse health literacy skills. Cancer. 2019 Jun 15;125(12):2066-2075. doi: 10.1002/cncr.31991. Epub 2019 Feb 27. PMID 30811591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: New lung, gastric and pancreatic cancer patients presenting to the University of Chicago outpatient oncology clinics, a large research institution located on Chicago's Southside, were identified for study accrual, using the electronic scheduling system.
Period: Overall Study
Arm/Group | Touchscreen Participants
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Touchscreen Participants: Testing Interactive Technology
Arm/Group | Touchscreen Participants
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants] — Self-reported age
  Participants
    <=18 years | 0
    Between 18 and 65 years | 99
    >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 116
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 96
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120
Clinical Trials Attitudes, Knowledge, and Interest [Mean (Full Range); unit: units on a scale] — Patients used the TT to self-administer 24 items from the Clinical Trial questionnaire developed by Jacobsen and colleagues measuring Receptivity (range: 1-5), Willingness (range: 1-5), Knowledge about cancer clinical trials (range:0-6), Positive Attitudes toward clinical trials (range:1-5), and Self-Efficacy (range: 1-5). A high score for each subscale represents a more favorable outcome.
  units on a scale
    Receptivity | 4.7 [2 to 5]
    Willingness | 4.1 [3 to 5]
    Knowledge | 3.3 [0 to 6]
    Positive Attitudes | 3.6 [2.6 to 5]
    Self-efficacy | 4.1 [2.3 to 5]
PROMIS [Mean (Standard Deviation); unit: T-score] — PROMIS Companionship Short Form, v2.0 - 6 items. PROMIS Instrumental Support Short Form, v2.0 - 6 items. PROMIS Global Health, v1.1 - 10 items assess overall health status (2 subscales: physical and mental health).
  All PROMIS measures are standardized so that a score of 50 (standard deviation of 10) represents the mean (and standard deviation) of the general U.S. population. A higher score denotes more support or better health.
  T-score
    Companionship | 56.4 (7.2)
    Instrumental Support | 59.5 (6.8)
    Physical Health | 48.4 (7.6)
    Mental Health | 46.1 (10.2)
Health Literacy [Mean (Standard Deviation); unit: t-score] — Health LiTT - The Health Literacy Assessment Using Talking Touchscreen Technology (Health LiTT) is a novel, self-administered multi-media test that meets psychometric standards (reliability of 0.90 or higher) for measurement of individual respondents, especially in the low to middle range of health literacy. Scores are standardized so that 50 (10) represents the mean (standard deviation) of the validation sample. A high score indicates better/high health literacy.
  t-score | 59.2 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Trials Attitudes, Knowledge, and Interest
Description: We hypothesized that our interactive educational tool would improve patient receptivity, willingness, knowledge, self-efficacy and positive attitudes regarding therapeutic cancer clinical trials through the use of patient-friendly technology in the immediate pre-visit period. Patients used the TT to self-administer 24 items from the Clinical Trial questionnaire developed by Jacobsen and colleagues measuring Receptivity (range: 1-5), Willingness (range: 1-5), Knowledge about cancer clinical trials (range: 0-6), Positive Attitudes toward clinical trials (range: 1-5), and Self-Efficacy (range: 1-5). A high score for each subscale represents a more favorable outcome.
Time Frame: Immediately after the visit.
Population: New lung, gastric and pancreatic cancer patients.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Touchscreen Participants
Number analyzed (Participants) | 120
units on a scale
  Receptivity | 4.6 [3 to 5]
  Willingness | 3.9 [2 to 5]
  Knowledge | 4.9 [1 to 6]
  Positive Attitude | 3.7 [2.6 to 4.9]
  Self-Efficacy | 4.3 [3.5 to 5]
Statistical Analysis 1: Comparison: Touchscreen Participants; Test type: Superiority; p = .307, t-test, 2 sided — This is for the receptivity sub-scale, and the comparison between pre and post-test scores; This was a paired t-test
Statistical Analysis 2: Comparison: Touchscreen Participants; Test type: Superiority; p = .009, t-test, 2 sided — This is for the willingness sub-scale, and the comparison between pre and posttest scores; This was a paired t-test
Statistical Analysis 3: Comparison: Touchscreen Participants; Test type: Superiority; p < .001, t-test, 2 sided — This is for knowledge sub scale, and the comparison between pre and posttest scores; A paired t-test
Statistical Analysis 4: Comparison: Touchscreen Participants; Test type: Superiority; p = .004, t-test, 2 sided — This is for the positive attitudes sub scale, and the comparison between pre and posttest scores; This was a paired t-test
Statistical Analysis 5: Comparison: Touchscreen Participants; Test type: Superiority; p < .001, t-test, 2 sided — This was for the self-efficacy sub scale, and the comparison between pre and posttest scores; This was a paired t-test

2. Secondary Outcome: Evaluate the Feasibility and Acceptability of Multi-media Technology.
Description: Secondary objectives of the study were to evaluate the feasibility and acceptability of multi-media technology for patient-reported outcomes (PRO) assessment and patient education in an oncology clinic. This was evaluated with a semi-structured interview with participants.
Time Frame: Immediately after the visit.
Population: A few people were not able to participate in the interviews.
Measure: Count of Participants; unit: Participants
Arm/Group | Touchscreen Participants
Number analyzed (Participants) | 109
Participants
  Difficulty using the touchscreen-not at all, a little bit | 102
  Overall rating of screen design-very good, excellent | 73
  Have you used a computer within the past 12 mo-yes | 98
  Have you ever used a touchscreen before-yes | 100
  Difficulty using the touchscreen to view the video or learning program-not at all | 99
  Overall rating of video-very good, excellent | 77
  Overall rating of learning program-very good, excellent | 78
  Did the video help you to better understand clinical trials-somewhat, quite a bit | 100
  Did the learning program (NC) help you to better understand clinical trials-somewhat, quite a bit | 94
  Overall rating of the amount of time you spent on this study, about right | 96
  Rate your experience participating-a little better, a lot better than expected | 61

3. Secondary Outcome: Clinical Trial Participation
Description: We used medical record abstraction to determine how many participants discussed clinical trials with their providers, how many were offered a clinical trial and how many were enrolled in a clinical trial.
Time Frame: About 6 months after the interview with participant.
Population: The percentages are based on the population described in the row titles.
Measure: Number; unit: Percentage of participants
Arm/Group | Touchscreen Participants
Number analyzed (Participants) | 120
Percentage of participants
  Discussed clinical trials with a physician | 63
  Offered a clinical trial among those who reported a discussion: number analyzed (Participants) | 76
  Offered a clinical trial among those who reported a discussion | 38
  Enrolled in a clinical trial among those offered a clinical trial: number analyzed (Participants) | 29
  Enrolled in a clinical trial among those offered a clinical trial | 48

ADVERSE EVENTS:
Time Frame: Not applicable to this study.
Description: Death and other serious and non-serious events were not collected.
Arm/Group | Touchscreen Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT02020252/Prot_SAP_000.pdf